CLINICAL TRIAL: NCT06344871
Title: Exploratory Study of NeuroLF, an Investigational Medical Device Without CE Marking for PET Imaging of the Human Brain
Brief Title: Exploratory Study Using a New Head-only PET Scanner / ExploreNeuroLF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Positrigo AG (Industry)
Collaborators: University of Zurich (Other); University of Leipzig (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 002
Record Dates: First submitted 2024-03-21; First posted 2024-04-03 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Brain Diseases
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NeuroLF Scan (Experimental): Scan on the NeuroLF PET system.
  Interventions: Device: NeuroLF
- Comparator Scan (Active Comparator): Scan on a conventional clinical PET system.
  Interventions: Device: Conventional PET scan

INTERVENTIONS:
Device: NeuroLF — NeuroLF Scan
  Arms: NeuroLF Scan
Device: Conventional PET scan — Scan on conventional PET system
  Arms: Comparator Scan

SUMMARY:
The "NeuroLF prototype" is a small aperture PET scanner. The NeuroLF prototype will be used with patients, which have just finished their regularly scheduled PET examination on a clinical whole body PET system. The radioactive tracer used for this procedure will still be active. This remaining acitivity will be used for an image acquisition with the NeuroLF prototype without the need for an additional radioactive tracer dose.

The control intervention is be a brain PET scan as part of standard clinical routine. It will be done immediately before the scan on the NeuroLF prototype.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving Informed Consent as documented by signature (Appendix Informed Consent Form).
* Ability to sit still in the head-only PET scanner for 15 minutes.
* Are scheduled to receive a regular brain PET scan as part of clinical routine.
* Male and Female patients 18 years to 80 years of age.

Exclusion Criteria:

* Contraindications to PET examination,
* Patient height smaller than 160 cm or taller than 200 cm,
* Patient weight more than 120 kg,
* Patient cannot sit upright for at least 15 minutes,
* Metal implants in the head,
* Pregnant or Breastfeeding women,
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug/device within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PET Image of the Brain | 1 day
  The primary outcome will be a PET image of the brain for each participant taken on NeuroLF. It will be compared against the image taken by the conventional PET machine by a trained physician and judged by whether it could be used for diagnosis and further analysis.

SECONDARY OUTCOMES:
Ease of Placement (Usability) | 1 day
  100-Visual Analog Scale question how easy it was to place the patient on NeuroLF vs. the comparator
Usage of accessories for patient placement (Usability) | 1 day
  Multiple Choice question which accessories were used to stabilize the patient.

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospital Leipzig, Leipzig, Germany
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No